CLINICAL TRIAL: NCT03268343
Title: A Phase 1 Open Label, Randomized, Two-Way Crossover Study in Healthy Volunteers to Investigate the Effect of Food on the Bioavailability of Cytisine
Brief Title: A Study in Healthy Volunteers to Investigate the Effect of Food on the Bioavailability of Cytisine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Achieve Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ACH-CYT-01; 2017-001562-19 (EudraCT Number)
Record Dates: First submitted 2017-08-25; First posted 2017-08-31 (Actual); Results first posted 2019-02-07 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — cytisine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Schedule A: Fed Then Fasted (Experimental): Schedule A (12 subjects):
  * Period 1: Cytisine (2 x 1.5 mg tablets) will be administered 30 minutes after the start of a high fat breakfast (fed state).
  * Period 2: Cytisine (2 x 1.5 mg tablets) will be administered after an overnight fast of at least 10 hours (fasting state).
  Interventions: Drug: Cytisine
- Schedule B: Fasted Then Fed (Experimental): Schedule B (12 subjects):
  * Period 1: Cytisine (2 x 1.5 mg tablets) will be administered after an overnight fast of at least 10 hours (fasting state).
  * Period 2: Cytisine (2 x 1.5 mg tablets) will be administered 30 minutes after the start of a high fat breakfast (fed state).
  Interventions: Drug: Cytisine

INTERVENTIONS:
Drug: Cytisine — Cytisine 1.5 mg Film-Coated Tablets
  Other Names: Tabex

SUMMARY:
This will be an open-label, randomised, 2-period, single-dose crossover study to determine the comparative bioavailability of cytisine following single-dose administration in healthy male and female subjects under fed and fasted conditions.

The study will be comprised of a pre-study screen, followed by 2 treatment periods (1 and 2) and a post-study follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males and females between 18 and 55 years of age.

   1. If a female subject of child bearing potential, a negative pregnancy test at screening and admission and willing to use an effective method of contraception (unless of non-childbearing potential or where abstaining from sexual intercourse is in line with the preferred and usual lifestyle of the subject) from first dose until 3 months after last dose of investigational medicinal product (IMP).
   2. If a female subject of non-child bearing potential, a negative pregnancy test at screening and admission. For the purposes of this study, this is defined as the subject being amenorrheic for at least 12 consecutive months or at least 4 months post-surgical sterilisation (including bilateral fallopian tube ligation or bilateral oophorectomy with or without hysterectomy). Menopausal status will be confirmed by demonstrating at screening that levels of follicle stimulating hormone (FSH) fall within the respective pathology reference range. In the event a subject's menopause status has been clearly established (for example, the subject indicates she has been amenorrheic for 10 years), but FSH levels are not consistent with a post-menopausal condition, determination of subject eligibility will be at Investigator's discretion following consultation with the Sponsor.
   3. If a male subject, willing to use an effective method of contraception (unless anatomically sterile or where abstaining from sexual intercourse is in line with the preferred and usual lifestyle of the subject) from first dose until 3 months after last dose of IMP.
2. Subject with a body mass index (BMI) of 18-32 kg/m^2. BMI = body weight in kg / [height in m]^2.
3. Subject with no clinically significant abnormal serum biochemistry, haematology and urine examination values within 28 days before the first dose of IMP.
4. Subject with negative urinary drugs of abuse screen, determined within 28 days before the first dose of IMP (a positive alcohol or cotinine result may be repeated at Investigator's discretion).
5. Subject with negative human immunodeficiency virus (HIV), hepatitis B surface antigen (Hep B) and hepatitis C virus antibody (Hep C) results.
6. Subject with no clinically significant abnormalities in 12-lead ECG determined after minimum of 5 minutes in supine position within 28 days before the first dose of IMP.
7. Subject with no clinically significant abnormalities in vital signs (systolic blood pressure between 90-150 mmHg, diastolic blood pressure (DBP) between 50 and 90 mmHg, and pulse rate (PR) between 40-110 bpm, measured on the dominant arm after minimum of 5 minutes in supine position) determined within 28 days before first dose of IMP.
8. Subject must be available to complete the study (including post study follow-up) and comply with study restrictions.
9. Subject must provide written informed consent to participate in the study.

Exclusion Criteria:

1. Known hypersensitivity/allergy reaction to varenicline, other cytisine-derivatives or any of the excipients in the Tabex formulation (lactose, cellulose, talc, magnesium).
2. History of severe hypersensitivity reactions to any other drugs.
3. History of any medical condition (e.g. gastrointestinal, renal or hepatic) or surgical condition (e.g. cholecystectomy, gastrectomy) that may affect drug pharmacokinetics (absorption, distribution, metabolism or excretion).
4. Difficulty in donating blood on either arm or known history.
5. History of alcoholism or drug abuse within last 2 years.
6. Regular nicotine intake (e.g., smoking, nicotine patch, nicotine chewing gum or electronic cigarettes) within previous 3 months and inability to refrain from nicotine intake from Screening until end of study.
7. Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements within 14 days (or 5 half-lives, whichever is longer) prior to the first dose of IMP, unless in the opinion of the Investigator the medication will not interfere with the study procedures or compromise subject safety.
8. Participated in any investigational drug clinical trial within the previous 3 months or a marketed drug trial within the previous 30 days prior to randomization on Day 1 of Period 1.
9. Donation of 450 mL or more blood or had history of significant blood loss due to any reason or had plasmapheresis within 3 months before the first dose of IMP.
10. Any special food restrictions that may hinder ability to consume the high fat breakfast provided during the study; such as lactose intolerance, vegan, low-fat, low sodium, etc.
11. Any inability or difficulty in fasting.
12. Inability to communicate well with Investigators (i.e., language problem, poor mental development or impaired cerebral function).
13. Any other condition that the Principal Investigator considers making the subject unsuitable for this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2017-08-08 (Actual); Primary Completion 2017-08-26 (Actual); Study Completion 2017-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Annelize Koch, MD, Principal Investigator — Simbec Research Ltd (Simbec)
Locations (1):
- Simbec Research Ltd, Merthyr Tydfil, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- 3 mg Cytisine, Schedule A: Fed Then Fasted: * Period 1: Cytisine (2 x 1.5 mg tablets) administered 30 minutes after the start of a high fat breakfast (fed state).
  * Period 2: Cytisine (2 x 1.5 mg tablets) administered after an overnight fast of at least 10 hours (fasting state).
- 3 mg Cytisine, Schedule B: Fasted Then Fed: * Period 1: Cytisine (2 x 1.5 mg tablets) administered after an overnight fast of at least 10 hours (fasting state).
  * Period 2: Cytisine (2 x 1.5 mg tablets) administered 30 minutes after the start of a high fat breakfast (fed state).
Period: Overall Study
Arm/Group | 3 mg Cytisine, Schedule A: Fed Then Fasted | 3 mg Cytisine, Schedule B: Fasted Then Fed
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- 3 mg Cytisine: 3 mg Cytisine, Schedule A: Fed Then Fasted
  * Period 1: Cytisine (2 x 1.5 mg tablets) administered 30 minutes after the start of a high fat breakfast (fed state).
  * Period 2: Cytisine (2 x 1.5 mg tablets) administered after an overnight fast of at least 10 hours (fasting state).
    3 mg Cytisine, Schedule B: Fasted Then Fed
  * Period 1: Cytisine (2 x 1.5 mg tablets) administered after an overnight fast of at least 10 hours (fasting state).
  * Period 2: Cytisine (2 x 1.5 mg tablets) administered 30 minutes after the start of a high fat breakfast (fed state).
Arm/Group | 3 mg Cytisine
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.1 (10.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 23
  Other, Not Specified | 1

OUTCOME MEASURES:

1. Primary Outcome: Plasma Cytisine Pharmacokinetics (PK): Maximum Observed Plasma Concentration (Cmax)
Time Frame: Pre-dose (within 60 minutes of dosing); 15 minutes, 20 minutes, 30 minutes, 45 minutes, 1 hour, 1.5 hours, 2 hours, 2.5 hours, 3 hours, 4 hours, 6 hours, 8 hours, 12 hours, 14 hours, 16 hours and 24 hours post-dose (+/- 1 minute)
Population: PK Set: All participants who received doses under both fed and fasted conditions and did not have an occurrence of vomiting which rendered the concentration profile unreliable. (Two participants were excluded for vomiting before twice the median Tmax had been reached following 3 mg cytisine administered in a fed state.)
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- 3 mg Cytisine, Fed: Cytisine (2 x 1.5 mg tablets) administered 30 minutes after the start of a high fat breakfast (fed state).
- 3 mg Cytisine, Fasted: Cytisine (2 x 1.5 mg tablets) administered after an overnight fast of at least 10 hours (fasting state).
Arm/Group | 3 mg Cytisine, Fed | 3 mg Cytisine, Fasted
Number analyzed (Participants) | 22 | 22
ng/mL | 22.9 (5.44) | 30.8 (7.91)
Statistical Analysis 1: Comparison: 3 mg Cytisine, Fed vs 3 mg Cytisine, Fasted; Test type: Superiority; Geometric LS Mean Ratio (%) = 74.71, 90% CI 2-sided [66.39 to 84.08] — fed / fasted; results obtained using an ANOVA with fixed effects of treatment, period, sequence and participant (sequence)

2. Primary Outcome: Plasma Cytisine PK: Total Area Under the Curve From Time Zero to Infinity (AUC0-∞)
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | 3 mg Cytisine, Fed | 3 mg Cytisine, Fasted
Number analyzed (Participants) | 22 | 22
h*ng/mL | 170 (30.3) | 176 (33.1)
Statistical Analysis 1: Comparison: 3 mg Cytisine, Fed vs 3 mg Cytisine, Fasted; Test type: Superiority; Geometric LS Mean Ratio (%) = 97.04, 90% CI 2-sided [94.20 to 99.98] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Plasma Cytisine PK: Time of Occurrence of Cmax (Tmax)
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | 3 mg Cytisine, Fed | 3 mg Cytisine, Fasted
Number analyzed (Participants) | 22 | 22
hours | 2.75 [0.500 to 6.12] | 0.75 [0.333 to 3.00]
Statistical Analysis 1: Comparison: 3 mg Cytisine, Fed vs 3 mg Cytisine, Fasted; Test type: Superiority; p < 0.0001, Wilcoxon Signed-Rank test; Median Difference (Final Values) = 1.38, 95% CI 2-sided [0.50 to 2.25] — Hodges-Lehmann method

4. Secondary Outcome: Plasma Cytisine PK: AUC From Time Zero to the Last Sampling Time (AUC0-t)
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | 3 mg Cytisine, Fed | 3 mg Cytisine, Fasted
Number analyzed (Participants) | 22 | 22
h*ng/mL | 163 (29.4) | 169 (33.0)
Statistical Analysis 1: Comparison: 3 mg Cytisine, Fed vs 3 mg Cytisine, Fasted; Test type: Superiority; Geometric LS Mean Ratio (%) = 96.52, 90% CI 2-sided [93.30 to 99.85] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Plasma Cytisine PK: Residual Area, or Percentage of Extrapolated Part for the Calculation of AUC0-∞ (AUC%)
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of extrapolated part
Arm/Group | 3 mg Cytisine, Fed | 3 mg Cytisine, Fasted
Number analyzed (Participants) | 22 | 22
percentage of extrapolated part | 4.37 (1.40) | 3.85 (1.46)

6. Secondary Outcome: Plasma Cytisine PK: Apparent Terminal Elimination Rate Constant (Lambda z)
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: 1/hour
Arm/Group | 3 mg Cytisine, Fed | 3 mg Cytisine, Fasted
Number analyzed (Participants) | 22 | 22
1/hour | 0.154 (0.0391) | 0.156 (0.0314)

7. Secondary Outcome: Plasma Cytisine PK: Apparent Terminal Elimination Half-Life (t1/2)
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | 3 mg Cytisine, Fed | 3 mg Cytisine, Fasted
Number analyzed (Participants) | 22 | 22
hours | 4.77 (1.16) | 4.59 (0.832)

8. Secondary Outcome: Urine Cytisine PK: Amount Excreted in Urine Over Time (Ae)
Time Frame: Pre-dose (within 30 minutes prior to first dose); 0-2 hours, 2-4 hours, 4-8 hours, 8-12 hours and 12-24 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | 3 mg Cytisine, Fed | 3 mg Cytisine, Fasted
Number analyzed (Participants) | 22 | 22
mg | 2.59 (0.407) | 2.47 (0.357)
Statistical Analysis 1: Comparison: 3 mg Cytisine, Fed vs 3 mg Cytisine, Fasted; Test type: Superiority; Geometric LS Mean Ratio (%) = 104.75, 95% CI 2-sided [98.97 to 110.87] — [estimate comment as in outcome 1, analysis 1]

9. Secondary Outcome: Urine Cytisine PK: Percentage of Drug Excreted in Urine (Ae%)
Description: To assess the renal elimination of cytisine via measurement of urinary concentrations of cytisine.
Time Frame: Pre-dose (within 30 minutes prior to first dose); 0-2 hours, 2-4 hours, 4-8 hours, 8-12 hours and 12-24 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of drug excreted
Arm/Group | 3 mg Cytisine, Fed | 3 mg Cytisine, Fasted
Number analyzed (Participants) | 22 | 22
percentage of drug excreted | 86.5 (13.6) | 82.4 (11.9)

10. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Serious TEAEs, and Discontinuation of Study Drug Due to AEs, by Severity and Relationship
Description: An adverse event (AE) is defined as any untoward medical occurrence which does not necessarily have a causal relationship with the treatment. TEAEs are defined as AEs not present prior to first administration of investigational product, or AEs present before first administration of study drug that worsen after the subject receives the first dose of study drug. A serious adverse event (SAE) is defined as an AE that: results in death; is life-threatening; requires hospitalization or prolongs existing inpatient's hospitalization; results in persistent or significant disability or incapacity; results in a congenital abnormality or birth defect; is an important medical event which requires medical intervention to prevent any of the above outcomes. Event severity was categorized as mild, moderate, or severe. Relationship of event to study drug was categorized as definite, probably, possible, unlikely, not related, or not applicable (N/A).
Time Frame: Day -1 to Day 7 plus 6-8 days (post-study follow-up)
Population: Safety Analysis Set: all participants who received at least one dose of cytisine.
Measure: Number; unit: participants
Arm/Group | 3 mg Cytisine, Fed | 3 mg Cytisine, Fasted
Number analyzed (Participants) | 24 | 24
participants
  ≥ 1 TEAE | 6 | 7
  ≥ 1 Serious TEAE | 0 | 0
  ≥ 1 TEAE Leading to Withdrawal of Study Drug | 0 | 0
  ≥ 1 Mild TEAE | 6 | 7
  ≥ 1 Moderate TEAE | 0 | 0
  ≥ 1 Severe TEAE | 0 | 0
  ≥ 1 TEAE Definitely Related to Study Drug | 0 | 0
  ≥ 1 TEAE Probably Related to Study Drug | 1 | 1
  ≥ 1 TEAE Possibly Related to Study Drug | 3 | 5
  ≥ 1 TEAE Unlikely Related to Study Drug | 1 | 1
  ≥ 1 TEAE Not Related to Study Drug | 0 | 0
  ≥ 1 TEAE Relationship to Study Drug = N/A | 1 | 0

ADVERSE EVENTS:
Time Frame: Day -1 to Day 7 plus 6-8 days (post-study follow-up)
Description: For each reporting group, a participant was counted only once per system organ class and preferred term. Consequently, if the same preferred term was observed for a participant in both fed and fasted states, the participant was counted only once in the "3 mg Cytisine, Overall" reporting group for that preferred term.
Groups:
- 3 mg Cytisine, Overall: Cytisine (2 x 1.5 mg tablets) administered 30 minutes after the start of a high fat breakfast (fed state).
  Cytisine (2 x 1.5 mg tablets) administered after an overnight fast of at least 10 hours (fasting state).
Arm/Group | 3 mg Cytisine, Fed | 3 mg Cytisine, Fasted | 3 mg Cytisine, Overall
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 6/24 | 7/24 | 10/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 3 mg Cytisine, Fed (N=24) | 3 mg Cytisine, Fasted (N=24) | 3 mg Cytisine, Overall (N=24)
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 1 | 2
Vomiting (Gastrointestinal disorders) | 2 | 1 | 3
Feeling hot (General disorders) | 0 | 1 | 1
Rhinitis (Infections and infestations) | 1 | 0 | 1
Dizziness (Nervous system disorders) | 2 | 3 | 4
Headache (Nervous system disorders) | 2 | 2 | 3
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1 | 1
Cold sweat (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Tooth repair (Surgical and medical procedures) | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigators are bound by requirements outlined in their individual clinical trial agreements with regard to publication of trial results.

DOCUMENTS (2):
  • Study Protocol (2017-05-19): https://cdn.clinicaltrials.gov/large-docs/43/NCT03268343/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-23): https://cdn.clinicaltrials.gov/large-docs/43/NCT03268343/SAP_001.pdf